CLINICAL TRIAL: NCT00001064
Title: A Pilot Study of Immunization With HIV-1 Antigen Pulsed Allogenic Dendritic Cells in HIV-Infected Asymptomatic Patients With CD4+ T Cells > 350 Cells/mm3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: SPIRAT 1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 1995-04

CONDITIONS: HIV Infections
Keywords: HIV Antigens; Immunotherapy, Adoptive; Dendritic Cells
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Allogenic Dendritic Cells

SUMMARY:
To define the safety and efficacy of sibling-supplied, HIV antigen-pulsed dendritic cells in increasing the immune response in HIV-infected patients.

Dendritic cells are a type of white blood cell used by the body to fight infection. They are instrumental in presenting antigens (such as HIV antigens) to the body's immune system. Since dendritic cells are not functioning maximally in HIV-infected patients, infusion of dendritic cells from an HIV-negative sibling may enable the affected sibling's immune system to recognize foreign particles more readily and increase immune response against the virus.

DETAILED DESCRIPTION:
Dendritic cells are a type of white blood cell used by the body to fight infection. They are instrumental in presenting antigens (such as HIV antigens) to the body's immune system. Since dendritic cells are not functioning maximally in HIV-infected patients, infusion of dendritic cells from an HIV-negative sibling may enable the affected sibling's immune system to recognize foreign particles more readily and increase immune response against the virus.

Dendritic cells from an HIV-negative sibling are obtained and treated with various viral proteins (HIV vaccines) or immunomodulators. The treated dendritic cells are infused into the HIV-infected patient monthly for 6 months. Siblings must be able to donate on multiple occasions, and patients are followed every 2-4 weeks during the study. Patients are screened over 3 months prior to study entry.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HLA A2+.
* Same cell type as donor sibling.
* CD4 count > 350 cells/mm3.
* HIV asymptomatic status.
* No HIV antivirals during study.
* Normal labs and chest x-ray.

Donor siblings must have:

* HLA A2+.
* HIV negativity.
* Ability to donate cells on multiple occasions.
* Negative status for hepatitis B and C.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiviral therapy (unless CD4 count declines to < 350 cells/mm3).

Prior Medication:

Excluded:

* Antiviral therapy within 90 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Univ School of Medicine, Stanford, California, United States